CLINICAL TRIAL: NCT03075800
Title: Integration of Illness Management and Recovery Within ACT
Acronym: ACT+IMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Maria Monroe-DeVita, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40487-C
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Severe Mental Illness; Schizophrenia; Bipolar Disorder
Keywords: Assertive Community Treatment (ACT) Only; Assertive Community Treatment (ACT) + Illness Management and Recovery (IMR)
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder | interventions — Community Mental Health Services; Salvage Therapy

STUDY DESIGN:
Intervention Model Description: A pilot, cluster randomized controlled trial was conducted in which ACT teams were randomized to provide either IMR within ACT (ACT+IMR) or standard ACT treatment (ACT-only). The impact of ACT+IMR vs. ACT-only on illness management and recovery outcomes was based on assessments conducted on a subset of randomly selected clients from each team, conducted at baseline, six months, and one year. Randomization to ACT+IMR or ACT-only was stratified by state and by team size, resulting in one large team and one small team assigned to each condition in each state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assertive Community Treatment (ACT) - Only (No Intervention): ACT is a multidisciplinary, team-based approach to providing a range of treatment, rehabilitation, and support services to high-need, high-risk people with severe mental illness who tend not to use clinic-based services; most services are provided on an outreach basis (e.g., in the person's home) and services are available 24 /7(27).
- Assertive Community Treatment+Illness Management and Recovery (Experimental): IMR follows a manualized curriculum to help clients pursue personal recovery goals and to teach them information, strategies, and skills over 11 modules (e.g., using medications, coping with stress) to manage their psychiatric illness. IMR can be provided in individual or group formats. The integrated ACT+IMR model was developed and manualized prior to the start of this evaluation (27). The model incorporates the following key features: a) ACT staff provide IMR in office-based group and/or individual sessions in office or community settings; b) regular community follow-up by ACT staff to assist clients with practicing IMR skills and achieving their goals; c) regular communication within ACT team (e.g., during daily meetings) on IMR client goals and progress; and d) supervision and consultation on IMR within ACT.
  Interventions: Behavioral: Assertive Community Treatment (ACT) + Illness Management and Recovery (IMR)

INTERVENTIONS:
Behavioral: Assertive Community Treatment (ACT) + Illness Management and Recovery (IMR) — The integrated ACT+IMR model was developed and manualized prior to the start of this evaluation (27). The model incorporates the following key features: a) ACT staff provide IMR in office-based group and/or individual sessions in office or community settings; b) regular community follow-up by ACT staff to assist clients with practicing IMR skills and achieving their goals; c) regular communication within ACT team (e.g., during daily meetings) on IMR client goals and progress; and d) supervision and consultation on IMR within ACT.
  Other Names: ACT+IMR
  Arms: Assertive Community Treatment+Illness Management and Recovery

SUMMARY:
Integrating Illness Management and Recovery (IMR) into Assertive Community Treatment (ACT) has great promise for improving the symptomatic, functional, and recovery outcomes for people with Serious Mental Illness (SMI), especially those individuals who have the greatest needs. In addition to these positive consumer outcomes, system benefits may also accrue due to more rapid graduation of consumers from ACT (with IMR) programs to less intensive levels of care. However, before these benefits can be realized, research and development are needed to design and pilot test a treatment manual that is feasible and acceptable to consumers and staff for integrating IMR and ACT.

DETAILED DESCRIPTION:
Despite significant advances in pharmacological treatments, many individuals with severe mental illnesses (SMI) such as schizophrenia and bipolar disorder continue to experience significant impairments in crucial life areas such as employment, housing, social functioning, and daily living skills. In addition, many of these individuals have significant levels of psychotic, mood, or negative symptoms, and are prone to frequent relapses and re-hospitalizations. Psychosocial treatments are needed to improve illness management and functioning beyond the limited effects of medication. However, relatively few psychosocial evidence-based practices (EBPs) exist for people with SMI and only a small percentage of people who could benefit from these treatments actually receive them. At the federal level, the implementation and dissemination of EBPs for people with SMI is a major policy priority and research objective.

Assertive Community Treatment (ACT) Overview. ACT is one of five psychosocial treatments for people with SMI designated as an EBP by SAMHSA. Since its inception, ACT has grown from a single, experimental research treatment program to an essential element within the service continuum of most public mental health systems for people with SMI. ACT programs typically serve consumers with the most severe symptoms who have the greatest disability and support needs (e.g., high rates of homelessness and hospitalizations), and who are most difficult to engage and retain in standard outpatient programs.

Research on ACT is extensive, with more than 25 RCTs. Literature reviews consistently conclude that ACT is more effective than standard community mental health services with demonstrated effectiveness in reducing psychiatric hospitalizations, and improving community tenure, retention in treatment, and high consumer and family satisfaction with services. However, ACT is less effective at improving symptom management, social functioning, and other functional outcomes, and needs to be adapted to better facilitate recovery. ACT is cost-effective compared to standard case management and has been widely disseminated with more than 300 ACT programs in at least 41 states.

Illness Management and Recovery (IMR) Overview. The Illness Management and Recovery (IMR) program is well-suited for enhancing outcomes in those areas less effectively addressed by ACT: symptom management and community functioning. IMR is also one of five psychosocial EBPs identified by SAMHSA for adults with SMI. IMR programs have been widely implemented across the U.S. and other countries, and researchers have conducted a number of open clinical trials and quasi-experimental studies. Recently, three RCTs were conducted, supporting the effectiveness of group-based IMR implemented in outpatient mental health clinics and supported housing. These studies show significant positive outcomes with IMR, including symptom reduction, improved functioning, increased knowledge about mental illness, and progress toward personal recovery goals.

Although these positive results support the effectiveness of IMR, several gaps and limitations are apparent in this growing area of practice and research. First, although IMR has been implemented clinically with very symptomatic consumers, such as inpatient and residential settings, controlled research on IMR has focused on outpatient settings, involving consumers who tend to be less symptomatic and higher functioning than those typically served on ACT teams. Second, providing IMR in outpatient clinics restricts the ability of clinicians to teach consumers skills in more natural community venues, which could improve the acquisition of new skills and related functional gains. Third, research on IMR has been mainly limited to the group modality, and hence, little is known about the effects of IMR provided in both individual and group formats.

Integrating IMR with ACT. Several characteristics of ACT suggest it will be an excellent platform for integrating and implementing the IMR program. By design, ACT programs serve people with the greatest needs who tend to drop out of standard outpatient programs; thus, integrating IMR into ACT has the potential to improve illness self-management in those consumers who need it most. The individualized and assertive outreach nature of ACT services will also allow IMR to be delivered in both individual and group modalities, and the in vivo practice of ACT will empower consumers to learn and practice IMR skills in their natural settings. Finally, the ACT principle of working with families and natural supports will facilitate the involvement of those supports in helping consumers to better manage their SMI and to achieve their recovery goals.

IMR also serves as an important potential service partner for ACT. ACT has been criticized by some as not being recovery-oriented. The integration of IMR may further enhance the growing recovery philosophy of ACT teams by providing a specific approach to promoting illness self-management and recovery that can be integrated into routine services. IMR can also improve the limited effectiveness of ACT teams at reducing symptoms and improving social and independent functioning. We also speculate (and plan to test in the subsequent, larger R01 research program) that providing IMR will accelerate the graduation of consumers from ACT, thereby increasing the number of slots available for new consumers in need of this scarce resource, further enhancing its cost-effectiveness. Thus, the integration of ACT and IMR has the potential to significantly benefit consumers with SMI, and increase the efficiency of the ACT model.

Despite these potential benefits, there are substantial challenges to integrating IMR into ACT teams. IMR has been developed and used primarily in traditional treatment settings, not in mobile community treatment approaches (e.g. ACT). In practice, many ACT clinicians find that their time is devoted to responding to daily crises and acute case management needs; ACT staff members often have difficulty making time and learning how to implement more learning-based and recovery-oriented interventions. Most critically, there are no standardized guidelines for implementing IMR within ACT, making the integration of the two EBPs even more challenging.

A few ACT teams, however, have foreseen the promise of integrating IMR into ACT. Using a nonequivalent group design, Garfinkle and Storch found that ACT consumers in IMR treatment showed a number of positive outcomes compared to ACT consumers without IMR services over 11 months, including lower hospitalization rates, improved retention of housing and competitive employment, and more work toward personal recovery goals. Salyers and colleagues conducted a small single group, pre-post pilot study to evaluate the feasibility of using peer specialists trained in IMR on ACT teams, and found that consumers who received IMR improved significantly on a measure of recovery, with a trend toward increased knowledge of mental illness, and consumer and staff satisfaction with IMR services. In a second study, Salyers and colleagues randomly assigned two of four ACT teams to IMR training and services (using only peer and mental health specialist staff for IMR service delivery). They reported that over the two-year period, ACT+IMR teams achieved moderate fidelity to IMR, but that rates of penetration were low, with only 25% of consumers having any exposure to IMR. However, secondary analyses found that ACT consumers who received IMR showed significant reductions in hospitalizations and incarcerations, and improvements in illness self-management.

The lack of well developed guidelines for implementing IMR undoubtedly limited the effectiveness of the program in the Salyers' project. Fortunately, lessons learned from this study, as well as the SAMHSA EBP study on IMR and the present project team's practice and research experience with both ACT and IMR, suggest that with a number of adaptations IMR can be successfully integrated into ACT services. We plan to develop and implement the following promising strategies for integrating these two EBPs in this project: (1) develop an adapted manual, training resources, and fidelity scale specific to implementing IMR within ACT, (2) provide intensive initial and follow-up booster clinician training, (3) provide regularly scheduled clinical supervision of IMR within the ACT team, in addition to regularly scheduled outside consultation by IMR+ACT experts during project startup, (4) create an organizational culture that supports and champions the integration of IMR within ACT, (5) cross-train all ACT staff to support the consumer's participation in IMR, and (6) create several specific, strategic adaptations to ACT team operations and protocol to facilitate the practice of IMR within daily ACT service activities. We expect these implementation strategies to result in an integrated IMR+ACT program that yields positive outcomes both to consumers and mental health service delivery systems.

ELIGIBILITY:
Eight ACT teams in two states were recruited, with four teams in each state.

Selection criteria included:

1. no prior IMR training; and
2. good fidelity to ACT, defined as a score > 3.5 (out of 5.0) on the Tool for Measurement of Assertive Community Treatment during state-sponsored fidelity assessments in 2012.

Ages: 23 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Illness Self-Management - The Clinician and Client Versions of the IMR Scale | baseline, 6, and 12 months
  evaluate illness self-management across 15 items rated on 5-point behaviorally anchored scales, with higher scores indicating better illness management. Overall scores are averages of the 15 items (ranging from 15 to 75).

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | baseline, 6, and 12 months
  Mental Health Symptoms
Daily Living Activities Scale (DLA-20), the Global Assessment of Functioning (GAF), and the Quality of Life Scale-Abbreviated (QLSA) | baseline, 6, and 12 months
  Psychosocial Functioning
Recovery Assessment Scale (RAS) | baseline, 6, and 12 months
  Recovery
Community Integration Measure (CIM) | baseline, 6, and 12 months
  Community Integration
Emergency mental health services | baseline, 6, and 12 months
  We examined two intensive services: emergency room and hospital admissions for mental health reasons. Research staff collected these data from ACT program staff for the 12-month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Monroe-DeVita, PhD, Principal Investigator — Co-PI, University of Washington, Seattle, WA; Gary Morse, PhD, Principal Investigator — Co-PI, Places for People, St. Louis, MO

IPD SHARING:
Plan to Share IPD: No